CLINICAL TRIAL: NCT02298712
Title: Biomarker for Hurler Disease - An International, Multicenter, Epidemiological Protocol
Brief Title: Biomarker for Hurler Disease (BioHurler)
Acronym: BioHurler
Status: Withdrawn | Type: Observational
Why Stopped: Transition to BioMetabol
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BHUR 06-2018
Record Dates: First submitted 2014-10-23; First posted 2014-11-24 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Mucopolysaccharidosis Type I; Gargoylism; Metabolism, Inborn Errors
Keywords: Iduronidase; Lysosomal Storage Diseases; Genetic Diseases, Inborn; Biomarker; Hurler-Scheie Syndrome; MPS I
MeSH Terms: conditions — Mucopolysaccharidosis I; Metabolism, Inborn Errors; Lysosomal Storage Diseases; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Laboratory Blood Test
  For the development of the new biomarkers using the technique of Mass-spectometry, a blood sample of maximal 10 ml blood will be taken via using a dry blood spot filter card. To proof the correct MPS1 diagnosis in those patients where up to the enrolment in the study no genetic testing has been done, sequencing of MPS1 will be done. The analyses will be done at the Centogene AG Am Strande 7 18055 Rostock Germany
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Patients with Hurler disease or high-grade suspicion for Hurler disease

SUMMARY:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Hurler disease from plasma. Testing for clinical robustness, specificity and long-term stability of the biomarker.

DETAILED DESCRIPTION:
Hurler disease - MPS I- (mucopolysaccharidosis I) is an inherited lysosomal storage disorder caused by a deficiency of alpha-L-iduronidase, a lysosomal enzyme normally required for the breakdown of certain complex carbohydrates known as glycosaminoglycans (GAGs). If the enzyme is not present in sufficient quantities, the normal breakdown of GAGs is incomplete or blocked. The cell is then unable to excrete the carbohydrate residues and they accumulate in the lysosomes of the cell. This accumulation disrupts the cell's normal functioning and gives rise to the clinical manifestations of the disease.

The incidence of MPS I is estimated to be at about 1 in 100,000 births. It is inherited in an autosomal recessive manner, affects males and females equally, and in most cases, both parents of an affected child are asymptomatic carriers of the disease. Types of MPS I. Children diagnosed with MPS I have historically been classified into one of three categories based on the severity of their symptoms and rate of disease progression. It has now become clear, however, that there is a wide spectrum of severity in MPS I with much overlap between the categories.

• Hurler Syndrome: The most severe form of MPS I is characterized by progressive developmental delay and severe progressive physical problems. Death often occurs before 10 years of age.

• Hurler-Scheie Syndrome: The intermediate form of MPS I is characterized by normal or near normal intelligence but more severe physical symptoms than those with Scheie Syndrome.

• Scheie Syndrome: The attenuated form of MPS I is characterized by normal intelligence, usually normal height, and milder physical problems than Hurler-Scheie. These individuals potentially have a normal life span.

Patients present within the first year of life with musculoskeletal alterations including short stature, dysostosis multiplex, thoracic-lumbar kyphosis, progressive coarsening of the facial features including large head with bulging frontal bones, depressed nasal bridge with broad nasal tip and anteverted nostrils, full cheeks and enlarged lips, cardiomyopathy and valvular abnormalities, neurosensorial hearing loss, enlarged tonsils and adenoids, and nasal secretion. Developmental delay is usually observed between 12 and 24 months of life and is primarily in the speech realm with progressive cognitive and sensorial deterioration. Hydrocephaly can occur after the age of two. Diffuse corneal compromise leading to corneal opacity becomes detectable from three years of age. Other manifestations include organomegaly, hernias and hirsutism. MPS1 syndrome is caused by mutations in the IDUA gene (4p16.3) leading to complete deficiency in the alpha-L-iduronidase enzyme and lysosomal accumulation of dermatan sulfate and heparan sulfate. Transmission is autosomal recessive. Early diagnosis is difficult because the first clinical signs are not specific, but it is very important to allow early treatment. Diagnosis is based on detection of increased urinary excretion of heparan and dermatan sulfate by 1, 9-dimethylmethylene blue (DMB) test and glycosaminoglycan (GAG) electrophoresis, and demonstration of enzymatic deficiency in leukocytes or fibroblasts. Genetic testing is available. Differential diagnoses include the milder form of mucopolysaccharidosis type 1, the MPS1-Scheie syndrome, although this form is associated with developmental delay with only slight cognitive impairment.

New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood (plasma) of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity.

Therefore it is the goal of the study to identify and validate a new biochemical marker from the plasma of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment.

Though MPS1 disease is a pan-ethnic disorder, the prevalence of this autosomal-recessive disorder is elevated in countries with a higher frequency of consanguinity. Therefore, we estimate that every 400th newborn in Arabian countries may be eligible for inclusion due to high-grade suspicion of MPS1 disease, while approximately every 2000th newborn in a non-Arabian country may be eligible.

ELIGIBILITY:
INCLUSION CRITERIA

* Informed consent will be obtained from the parents before any study related procedures.
* Patients of both gender older than 2 month
* The patient has a diagnosis of Hurler disease or a high-grade suspicion for Hurler disease
* High-grade suspicion present, if one or more inclusion criteria are valid:

  1. - Positive family anamnesis for Hurler disease
  2. - Macrocephaly
  3. - Deformed bones and stiff joints, especially the spine, hips, knees, wrists and fingers
  4. - Musculoskeletal alterations including short stature
  5. - Developmental delay and/or progressive mental deterioration

EXCLUSION CRITERIA

* No Informed consent from the parents before any study related procedures.
* Patients of both gender younger than 2 month
* No diagnosis of Hurler disease or no valid criteria for profound suspicion of Hurler disease

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Hurler disease or high-grade suspicion for Hurler disease
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Hurler disease from blood | 24 months
  New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity.

SECONDARY OUTCOMES:
Testing for clinical robustness, specificity and long-term stability of the biomarker | 36 months
  the goal of the study to identify and validate a new biochemical marker from the blood of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Study Chair — Centogene GmbH
Locations (5):
- Children's Hospital, Faculty of Medicine, Ain Shams University, Cairo, Egypt
- Centogene AG, Rostock, Germany
- India (2):
  - Amrita Institute of Medical Sciences & Research Centre, Kochi, Kerala
  - Navi Mumbai Institute of Research In Mental And Neurological Handicap (NIRMAN), Mumbai
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: Undecided